CLINICAL TRIAL: NCT00391807
Title: Open-Label Study of the Safety and Efficacy of a Low Dose Oral Contraceptive Containing Norethindrone Acetate and Ethinyl Estradiol
Brief Title: Study of Safety and Efficacy of an Oral Contraceptive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-05806
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Contraception
Keywords: Contraception
MeSH Terms: interventions — Norethindrone Acetate; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study drug (Experimental): Norethindrone/Ethinyl Estradiol
  Interventions: Drug: Norethindrone acetate/ethinyl estradiol

INTERVENTIONS:
Drug: Norethindrone acetate/ethinyl estradiol — one tablet per day

SUMMARY:
This is a non-comparative study. The primary objective of the study is to assess the efficacy of a low dose oral contraceptive in the prevention of pregnancy. The secondary objectives are to assess the incidence of intracyclic bleeding; and to assess the safety and tolerability of the product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Women
* Age 18-45
* At risk for pregnancy
* History of regular cycles

Exclusion Criteria:

* Contraindications for use of hormonal contraception
* Conditions which affect the absorption or metabolism of steroid hormones
* BMI > 35

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1683 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Sponsor GmbH
Locations (55):
- United States (55):
  - Warner Chilcott Investigational Site, Phoenix, Arizona
  - Warner Chilcott Investigational Site, Tempe, Arizona
  - Warner Chilcott Investigational Site, Tucson, Arizona
  - Warner Chilcott Investigational Site, Carmichael, California
  - Warner Chilcott Investigational Site, San Diego, California
  - Warner Chilcott Investigational Site, Denver, Colorado
  - Warner Chilcott Investigational Site, Boynton Beach, Florida
  - Warner Chilcott Investigational Site, Clearwater, Florida
  - Warner Chilcott Investigational Site, Jacksonville, Florida
  - Warner Chilcott Investigational Site, Leesburg, Florida
  - Warner Chilcott Investigational Site, Longwood, Florida
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, New Port Richey, Florida
  - Warner Chilcott Investigational Site, Pembroke Pines, Florida
  - Warner Chilcott Investigational Site, Plantation, Florida
  - Warner Chilcott Investigational Site, St. Petersburg, Florida
  - Warner Chilcott Investigational Site, West Palm Beach, Florida
  - Warner Chilcott Investigational Site, Roswell, Georgia
  - Warner Chilcott Investigational Site, Sandy Springs, Georgia
  - Warner Chilcott Investigational Site, Champaign, Illinois
  - Warner Chilcott Investigational Site, Peoria, Illinois
  - Warner Chilcott Investigational Site, Indianapolis, Indiana
  - Warner Chilcott Investigational Site, Wichita, Kansas
  - Warner Chilcott Investigational Site, Lexington, Kentucky
  - Warner Chilcott Investigational Site, Louisville, Kentucky
  - Warner Chilcott Investigational Site, Berlin, New Jersey
  - Warner Chilcott Investigational Site, Lawrenceville, New Jersey
  - Warner Chilcott Investigational Site, Moorestown, New Jersey
  - Warner Chilcott Investigational Site, Albuquerque, New Mexico
  - Warner Chilcott Investigational Site, Cary, North Carolina
  - Warner Chilcott Investigational Site, New Bern, North Carolina
  - Warner Chilcott Investigational Site, Raleigh, North Carolina
  - Warner Chilcott Investigational Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Site, Cleveland, Ohio
  - Warner Chilcott Investigational Site, Columbus, Ohio
  - Warner Chilcott Investigational Site, Oklahoma City, Oklahoma
  - Warner Chilcott Investigational Site, Portland, Oregon
  - Warner Chilcott Investigational Site, Philadelphia, Pennsylvania
  - Warner Chilcott Investigational Site, Pittsburgh, Pennsylvania
  - Warner Chilcott Investigational Site, Pottstown, Pennsylvania
  - Warner Chilcott Investigational Site, Charleston, South Carolina
  - Warner Chilcott Investigational Site, Columbia, South Carolina
  - Warner Chilcott Investigational Site, Greenville, South Carolina
  - Warner Chilcott Investigational Site, Dallas, Texas
  - Warner Chilcott Investigational Site, Houston, Texas
  - Warner Chilcott Investigational Site, San Antonio, Texas
  - Warner Chilcott Investigational Site, Magna, Utah
  - Warner Chilcott Investigational Site, Salt Lake City, Utah
  - Warner Chilcott Investigational Site, Sandy City, Utah
  - Warner Chilcott Investigational Site, Norfolk, Virginia
  - Warner Chilcott Investigational Site, Richmond, Virginia
  - Warner Chilcott Investigational Site, Virginia Beach, Virginia
  - Warner Chilcott Investigational Site, Seattle, Washington
  - Warner Chilcott Investigational Site, Spokane, Washington
  - Warner Chilcott Investigational Site, Tacoma, Washington

REFERENCES:
- [Derived] Nakajima ST, Pappadakis J, Archer DF. Body mass index does not affect the efficacy or bleeding profile during use of an ultra-low-dose combined oral contraceptive. Contraception. 2016 Jan;93(1):52-7. doi: 10.1016/j.contraception.2015.09.013. Epub 2015 Sep 26. PMID 26410176
- [Derived] Archer DF, Nakajima ST, Sawyer AT, Wentworth J, Trupin S, Koltun WD, Gilbert RD, Ellman H. Norethindrone acetate 1.0 milligram and ethinyl estradiol 10 micrograms as an ultra low-dose oral contraceptive. Obstet Gynecol. 2013 Sep;122(3):601-7. doi: 10.1097/AOG.0b013e3182a1741c. PMID 23921878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 01 Nov '06 thru 24 Aug '08
Groups:
- Norethindrone/Ethinyl Estradiol: 1 tablet norethindrone acetate (NETA) 1mg/ethinyl estradiol (EE)10 mcg daily for 24 days, 1 EE 10 mcg tablet daily for 2 days, 1 inactive ferrous fumarate tablet daily for 2 days
Period: Overall Study
Arm/Group | Norethindrone/Ethinyl Estradiol
Started | 1683
Completed | 968
Not Completed | 715
Not completed — Did not receive study medication | 23
Not completed — Adverse Event | 177
Not completed — Pregnancy | 25
Not completed — Lost to Follow-up | 227
Not completed — Withdrawal by Subject | 147
Not completed — Protocol Violation | 20
Not completed — Various | 96

BASELINE CHARACTERISTICS:
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1683
Age Continuous [Mean (Standard Deviation); unit: years] — MITT (Modified Intent to Treat) Population
  years | 28.6 (6.9)
Age, Customized [Number; unit: participants] — MITT Population
  participants
    18-35 years | 1295
    >35 years | 287
Gender [Number; unit: participants] — MITT Population
  participants
    Female | 1582
    Male | 0
Region of Enrollment [Number; unit: participants] — MITT Population
  participants
    United States | 1582

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate (Expressed as Pearl Index) in Women Aged 18 to 35, MITT Population,
Time Frame: 13 cycles, 28 days each (1 year)
Population: Modified Intent to Treat Population (MITT), Women Aged 18-35, 27 women had no cycles evaluable for pregnancy because they used alternative contraceptive methods in all cycles - 1555 subjects evaluable in MITT population. Number of pregnancies per 100 women-years of treatment in MITT Population
Measure: Number; unit: Pregnancy Rate
Units Other Than Participants: Pregnancies
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1266
Number analyzed (Pregnancies) | 24
Pregnancy Rate | 2.554

2. Secondary Outcome: Number of Intracyclic Bleeding (IB)/Spotting Days Cycle 2, MITT Population
Description: MITT Population
Time Frame: 2 Cycles, 28 days each (56 days)
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Bleeding/Spotting Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Bleeding/Spotting Days | 3.21 (4.15)

3. Primary Outcome: Pregnancy Rate (Expressed as Pearl Index) in Women Aged 18-45, MITT Population
Time Frame: 13 Cycles, 28 days each (1 year)
Population: MITT Population, All Subjects 18-45 years old, 27 women had no cycles evaluable for pregnancy because they used alternative contraceptive methods in all cycles - 1555 subjects evaluable in MITT population. Number of pregnancies per 100 women-years of treatment in MITT Population
Measure: Number; unit: Pregnancy Rate
Units Other Than Participants: Pregnancies
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1555
Number analyzed (Pregnancies) | 26
Pregnancy Rate | 2.167

4. Secondary Outcome: Number of Intracyclic Bleeding (IB)/Spotting Days Cycle 6, MITT Population
Description: MITT Population
Time Frame: 6 cycles, 28 days each (168 days)
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Bleeding/Spotting Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Bleeding/Spotting Days | 2.00 (3.12)

5. Secondary Outcome: Number of Intracyclic Bleeding (IB)/Spotting Days Cycle 13, MITT Population
Description: MITT Population
Time Frame: 13 cycles, 28 days each (1 year)
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Bleeding/Spotting Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Bleeding/Spotting Days | 1.81 (3.01)

6. Secondary Outcome: Percentage of Subjects With Withdrawal Bleeding (%), Cycle 2, MITT Population
Time Frame: 2 cycles, 28 days each (56 days)
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Percentage of Participants | 34.8

7. Secondary Outcome: Percentage of Subjects With Withdrawal Bleeding (%), Cycle 6, MITT Population
Time Frame: 6 cycles, 28 days each (168 days)
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Percentage of Participants | 25.0

8. Secondary Outcome: Percentage of Subjects With Withdrawal Bleeding (%), Cycle 13, MITT Population
Time Frame: 13 cycles, 28 days each (1 year)
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Percentage of Participants | 22.4

9. Secondary Outcome: Median Duration of Withdrawal Bleeding, Cycle 2, MITT Population
Time Frame: 2 cycles, 28 days each (56 days)
Population: MITT Population
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Days | 3.93 (2.18)

10. Secondary Outcome: Median Duration of Withdrawal Bleeding, Cycle 6, MITT Population
Time Frame: 6 cycles, 28 days each (168 days)
Population: MITT Population
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Days | 3.99 (2.11)

11. Secondary Outcome: Median Duration of Withdrawal Bleeding, Cycle 12, MITT Population
Time Frame: 12 cycles, 28 days each (336 days)
Population: MITT Population
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Days | 3.85 (2.07)

12. Secondary Outcome: Total Number of Bleeding Days Per Cycle, Cycle 2, MITT Population
Time Frame: 2 cycles, 28 days each (56 days)
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Days | 4.57 (4.94)

13. Secondary Outcome: Total Number of Bleeding Days Per Cycle, Cycle 6, MITT Population
Time Frame: 6 cycles, 28 days each (168 days)
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Days | 3.00 (3.73)

14. Secondary Outcome: Total Number of Bleeding Days Per Cycle, Cycle 13, MITT Population
Time Frame: 13 cycles, 28 days each (1 year)
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Days | 3.36 (4.51)

15. Secondary Outcome: Percentage of Subjects With Amenorrhea, Cycle 2, MITT Population
Time Frame: 2 cycles, 28 days each (56 days)
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Percentage of Participants | 30.7

16. Secondary Outcome: Percentage of Subjects With Amenorrhea, Cycle 6, MITT Population
Time Frame: 6 cycles, 28 days each (168 days)
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Percentage of Participants | 42.9

17. Secondary Outcome: Percentage of Subjects With Amenorrhea, Cycle 13, MITT Population
Time Frame: 13 cycles, 28 days each (1 year)
Population: MITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 1582
Percentage of Participants | 49.1

ADVERSE EVENTS:
Time Frame: 1 Nov 2006 thru 27 Aug 2008 - 1 year, 9 months
Description: 1683 Subjects Randomized but 23 subjects did not take study medication therefore 1660 subjects evaluated for adverse events.
Arm/Group | Norethindrone/Ethinyl Estradiol
Serious Adverse Events (participants affected / at risk) | 15/1660
Other Adverse Events (participants affected / at risk) | 390/1660
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norethindrone/Ethinyl Estradiol (N=1660)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3)
Hyperemesis Gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Venous Thrombosis (Ovarian) (Vascular disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1)
Transverse Sinus Thrombosis (Nervous system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Partial Hysterectomy with Bladder Sling (Elective Therapeutic Procedure) (Surgical and medical procedures) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norethindrone/Ethinyl Estradiol (N=1660)
Headache (Nervous system disorders) | 116 (116)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 103 (103)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 86 (86)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 85 (85)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less